CLINICAL TRIAL: NCT06713239
Title: A Randomized Comparison of Personalized Management for Medical and Interventional Therapy Based On Coronary Atherosclerotic Plaque Versus Usual Care for Symptomatic Patients With Suspicion of CAD
Brief Title: A Randomized Comparison of Personalized Therapy Mgmt Based On Coronary Atherosclerotic Plaque Vs. Usual Care for Symptomatic Patients With Suspicion of CAD
Acronym: PARAMOUNT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cleerly, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00082528
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Coronary Plaque-Based Care (Experimental): Patients randomized to the Coronary Plaque-Based Care arm will undergo CCTA with AI-enabled quantitative assessment of the morphology and composition of coronary atherosclerotic plaque and will receive medical and interventional management informed by CCTA findings and per discretion of the treating physician. All patients will receive a standardized assessment of clinical and risk factor status at baseline and 180 days.
  Interventions: Device: Cleerly Labs and Cleerly ISCHEMIA
- Usual Care (No Intervention): Patients randomized to the Usual Care arm will be referred to their usual care providers for standard of care management post stress test findings, possibly including coronary angiography and/or revascularization per the treating provider's recommendation. All patients will receive a standardized assessment of clinical and risk factor status at baseline and 180 days.

INTERVENTIONS:
Device: Cleerly Labs and Cleerly ISCHEMIA — Participants in the coronary plaque-based care arm will have CCTA at baseline. CCTA images will be redacted and uploaded to Cleerly, interpreted using Cleerly Labs and Cleerly ISCHEMIA, and archived.
  Arms: Coronary Plaque-Based Care

SUMMARY:
PARAMOUNT is a prospective randomized open-label trial testing the hypothesis that a personalized management strategy in symptomatic patients with suspicion of coronary artery disease (CAD), using a CT-based coronary atherosclerotic plaque assessment by AI-enabled quantitative software improves: certainty for diagnosis of CAD, control of CAD risk factors and efficiency of ICA referral with appropriate PCI compared to the usual care strategy based on current AHA/ACC guidelines for care of symptomatic patients with suspicion of CAD.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Symptomatic patients with suspicion of CAD, including those referred for elective, non-urgent diagnostic testing (e.g. stress test)

Exclusion Criteria:

* LDL < 100 mg/dL
* Currently or previously treated beyond primary prevention guidelines
* Suspected acute coronary syndrome or otherwise unstable clinical status
* Planned cardiovascular procedure (e.g. coronary angiography, cardiac surgery, non-coronary vascular procedure)
* Noninvasive or invasive CV testing for CAD within 1 year (e.g. invasive coronary angiography (ICA), coronary CT angiography (CCTA) including calcium scoring)
* Known history of obstructive CAD (prior myocardial infarction, CABG or PCI, stenosis ≥50%)
* Known EF ≤40% or other moderate to severe valvular or congenital cardiac disease
* Contraindications to CCTA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to determine whether a management strategy improves efficiency and effectiveness. | Through study completion- an average of 1 year
  The primary endpoint is composed of multuple elements, which are to be compared between Coronary Plaque-Based care and the usual care arm, in a hierarchical fashion, using the win ratio approach:
  1. Improved diagnostic certainty of CAD
The primary objective of this study is to determine whether a management strategy improves efficiency and effectiveness. | Through study completion- an average of 1 year
  The primary endpoint is composed of multuple elements, which are to be compared between Coronary Plaque-Based care and the usual care arm, in a hierarchical fashion, using the win ratio approach:
  2. Reduction in LDL
The primary objective of this study is to determine whether a management strategy improves efficiency and effectiveness. | Through study completion- an average of 1 year
  The primary endpoint is composed of multuple elements, which are to be compared between Coronary Plaque-Based care and the usual care arm, in a hierarchical fashion, using the win ratio approach:
  3. Freedom from ICA without a finding of obstructive CAD
The primary objective of this study is to determine whether a management strategy improves efficiency and effectiveness. | Through study completion- an average of 1 year
  The primary endpoint is composed of multuple elements, which are to be compared between Coronary Plaque-Based care and the usual care arm, in a hierarchical fashion, using the win ratio approach:
  4. Freedom from PCI without finding of clinically significant stenosis

SECONDARY OUTCOMES:
The secondary objective of the study is to determine whether a management strategy improves patients' experience of chest pain, quality of life, and adherence to medication. | Through study completion- an average of 1 year
  The secondary endpoints assess angina symptoms, medication adherence, and quality of life.
  1. Change in angina symptoms assessed using the Seattle Angina Questionnaire.
The secondary objective of the study is to determine whether a management strategy improves patients' experience of chest pain, quality of life, and adherence to medication. | Through study completion- an average of 1 year
  The secondary endpoints assess angina symptoms, medication adherence, and quality of life.
  2. Medication adherence assessed using the Voils DOSE-Nonadherence measure (Blalock, et al. 2019).
The secondary objective of the study is to determine whether a management strategy improves patients' experience of chest pain, quality of life, and adherence to medication. | Through study completion- an average of 1 year
  The secondary endpoints assess angina symptoms, medication adherence, and quality of life.
  3. Quality of life assessed using the 20-item Short Form Survey (SF-20).

CONTACTS AND LOCATIONS:
Overall Officials: Todd Villines, MD, Principal Investigator — University of Virginia; Maros Ferencik, MD, Principal Investigator — Oregon Health and Science University
Locations (21):
- United States (21):
  - Cardiology Associates of Mobile, Mobile, Alabama
  - Valiance Clinical Research- Huntington Park, Huntington Park, California
  - Cardiovascular Institute of San Diego, San Diego, California
  - Valiance Clinical Research- Tarzana, Tarzana, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Intermountain Health Saint Joseph Hospital, Broomfield, Colorado
  - Tampa Cardiovascular Interventions and Research, Tampa, Florida
  - Flourish Research, Winter Park, Florida
  - Endeavor Health Clinical Operations, Evanston, Illinois
  - MercyOne Des Moines Medical Center, West Des Moines, Iowa
  - Saint Elizabeth Medical Center, Edgewood, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Flourish- Bowie, Bowie, Maryland
  - St. Louis Heart and Vascular, Bridgeton, Missouri
  - Advanced Heart and Vascular Institute of Hunterdon, Flemington, New Jersey
  - Capital Cardiology Associates, Albany, New York
  - University of Cincinnatti, Cincinnati, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - The University of Tennessee Medical Center, Knoxville, Tennessee
  - Medical City Fort Worth Hospital, Fort Worth, Texas
  - Chippenham and Johnston Willis Hospitals, Richmond, Virginia